CLINICAL TRIAL: NCT02062762
Title: Internet-based Stress Reduction Training for Students - a Pilot Study
Brief Title: Internet-based Stress Reduction Training for Students
Acronym: IBSR-stud
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Richard Branstrom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KI-MBSR-Pilot
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Depression; Stress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online-MBSR (Experimental): 8 week mindfulness based stress reduction online
  Interventions: Behavioral: Online-MBSR
- Expressive Writing Online (Active Comparator): Online distributed expressive writing intervention as active control
  Interventions: Behavioral: Expressive Writing Online

INTERVENTIONS:
Behavioral: Online-MBSR — 8 week mindfulness based stress reduction online
  Arms: Online-MBSR
Behavioral: Expressive Writing Online — Online distributed expressive writing intervention as active control
  Arms: Expressive Writing Online

SUMMARY:
The main objective of the current study is to evaluate whether a mindfulness based intervention delivered online can provide an effective resource for increasing psychological well-being among students. In addition, explore potential mechanisms through which the training lead to improvements by means of mediational analyses, with hypothesized variables like positive/negative affect and attention regulation.

ELIGIBILITY:
Inclusion Criteria:

* current student
* have an active e-mail account
* regular use of the internet

Exclusion Criteria:

* non-Swedish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Psychological well-being | Baseline, Week 8
  Change over time

SECONDARY OUTCOMES:
Depression symptoms | Baseline, Week 8
  Change over time

OTHER OUTCOMES:
Health-related behaviors | Baseline, Week 8
  Change over time in proportion reporting binge drinking of alcohol past week (yes/no), and cigarette smoking past week (yes/no); both assessed though self-report questionnaire items.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Branstrom, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinsk Institute, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Kvillemo P, Brandberg Y, Branstrom R. Feasibility and Outcomes of an Internet-Based Mindfulness Training Program: A Pilot Randomized Controlled Trial. JMIR Ment Health. 2016 Jul 22;3(3):e33. doi: 10.2196/mental.5457. PMID 27450466